CLINICAL TRIAL: NCT05376202
Title: Fluorescent Guided Surgery in Penile Carcinoma Using Cetuximab-800IRDyeCW
Brief Title: Image Guided Penile Cancer Surgery
Acronym: GLANS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Max J.H. Witjes, Prof. dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 202000333
Record Dates: First submitted 2022-04-19; First posted 2022-05-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Penile Cancer; Margin Assessment
MeSH Terms: conditions — Penile Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 1: 75mg Cetuximab and 15mg Cetuximab-IRDye800CW (Experimental): Patients receive 75mg of Cetuximab, followed by 15mg Cetuximab-IRDye800CW I.V. two days prior to surgery.
  Interventions: Drug: Cetuximab-IRDye800CW

INTERVENTIONS:
Drug: Cetuximab-IRDye800CW — Patients will receive 75mg Cetuximab followed by 15mg Cetuximab-IRDye800CW two days prior to surgery

SUMMARY:
The main treatment modality for Penile Squamous Cell Carcinoma (PSCC) is surgery with curative intent. In organ sparing surgery a tumor-positive margin of up to 36% exist. Tumor-positive surgical margins are an independent risk factor for local recurrence, which has been reported to be up to 18%. Tumor-positive margins always lead to extra, penile sparing surgery, which leads to longer hospitalization, higher exposure to anesthetic interventions and a worse psychological outcome.

Currently, no intraoperative imaging technique that provides real time feedback for resection margins exists in PSCC. Molecular fluorescence-guided Surgery (MFGS) using targeted near-infrared (NIR) optical contrast agents like for example Cetuximab-800CW is a promising technique to accommodate this need. Epidermal Growth Factor Receptor (EGFR) is overexpressed in PSCC and has safely and successfully been used as target for molecular imaging, particularly for assessment for tumor margins in head and neck squamous cell carcinoma (ICON study, UMCG1).

DETAILED DESCRIPTION:
The main treatment modality for Penile Squamous Cell Carcinoma (PSCC) is surgery with curative intent. There is no difference in mortality between organ sparing surgery and radical surgery, and for optimal cosmetic and functional results small resection (3-5mm) margins are used. In organ sparing surgery a tumor-positive margin of up to 36% exist. Tumor-positive surgical margins are an independent risk factor for local recurrence, which has been reported to be up to 18%. These local remaining tumor depositions can be continuous or discontinuous from the main tumor, which makes it hard for the treating surgeon to recognize them clinically. Tumor-positive margins always lead to extra, penile sparing surgery, which leads to longer hospitalization, higher exposure to anesthetic interventions and a worse psychological outcome.

Currently, no intraoperative imaging technique that provides real time feedback for resection margins exists in PSCC. Molecular fluorescence-guided Surgery (MFGS) using targeted near-infrared (NIR) optical contrast agents like for example Cetuximab-800CW is a promising technique to accommodate this need. Epidermal Growth Factor Receptor (EGFR) is overexpressed in PSCC and has safely and successfully been used as target for molecular imaging, particularly for assessment for tumor margins in head and neck squamous cell carcinoma (ICON study, UMCG1).

Objectives:

The purpose of the current study is to determine the feasibility of using MFGS using Cetuximab-800CW as an intraoperative margin assessment tool for penile carcinoma.

Study design:

The study is a single-center prospective, phase1 feasibility study. In total, fifteen patients with biopsy proven PSCC will be included. 2-4 days before surgery, a predose of 75mg 'cold' cetuximab will be administered intravenously, followed by 15mg of cetuximab-800CW intravenously, with 1 hour between start of the cold dose and the cetuximab-800CW. After 3 patients are included, an interim analysis will be performed. If a tumor to background of >2 is obtained with either in vivo or ex-vivo analysis, the next 12 patients will be included. If a TBR of <2 is reached, the dose of cetuximab-800CW will be increased to 25mg with the same predosing scheme, 75mg of cold cetuximab. When 3 patients are included in the second dose group, a second interim analysis will be performed. If a tumor to background of >2 is obtained by ex-vivo analysis, 12 patients more will be included. If a TBR of <2 is found, the study will be terminated.

Study population:

Patients with histologically proven PSCC who meet all in- and exclusion criteria, and are opted for primary surgery as their treatment.

Patient related study procedures:

After written informed consent is obtained, patients will receive an intravenous administration of 75mg 'cold' cetuximab followed by 15mg of cetuximab-800CW 1 hour after the administration of the predose. 2-4 days after the injection of the imaging agent, fluorescence imaging is performed intraoperatively, both in vivo and ex vivo. 1 day after surgery, fluorescence imaging will again be performed during pathological processing on the excised tissue. Both intraoperatively and during the pathology process, fluorescence will be quantified by MDSFR/SFF spectroscopy.

Main study parameters/endpoints:

The main objective of this feasibility study is to investigate whether cetuximab-800CW could be used for margin assessment during surgery in patients with PSCC.

Burden, risks and benefit related to participation.

Burden:

The extra burden the patients associated with the study procedure is an extra visit to the hospital 2-4 days before surgery for the administration of cetuximab-800CW. This will take approximately 2 hours. Also, the surgical procedure will be prolonged 15-20 minutes due to fluorescence imaging and spectroscopy measurements.

Risks:

Risks to study participants are mainly related to the risks of the administration of the imaging agent. No preclinical or clinical study reported higher than grade 2 adverse events using cetuximab-800CW, moreover, these studies used significant higher doses of the investigational product. Previous studies with cetuximab-800CW reported no imaging agent related serious events. Currently, a phase 2 trial is performed at the UMCG with Cetuximab-800CW (NCT03134846), no grade 2 or higher imaging agent related serious advents were reported so far.

Benefit:

Patients will have no benefit from this study directly. Surgery will be planned as usual. During surgery, no decisions will be made based on the fluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed diagnosis of primary or recurrent PSCC and scheduled to undergo surgical resection of primary or recurrent tumor with or without (sentinel) lymph node procedure as decided by the Urology Department of the UMCG.
2. Age ≥ 18 years
3. Written informed consent
4. Adequate potential for follow-up

Exclusion Criteria:

1. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
2. Concurrent uncontrolled medical conditions
3. Received an investigational drug within 30 days prior to the dose of cetuximab-800CW
4. Tumors at sites of which the surgeon would assess that in vivo imaging would not be feasible
5. Had within 6 months prior to enrollment: myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease, unstable angina
6. Inadequately controlled hypertension with or without current antihypertensive medications
7. History of infusion reactions to cetuximab or other monoclonal antibody therapies
8. Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females)
9. Lab values that in the opinion of the primary surgeon would prevent surgical resection
10. Patients receiving Class Ia (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
11. Magnesium, potassium and calcium deviations that might lead to cardiac rhythm (grade II or higher deviations by CTCAE)
12. Life expectancy < 12 weeks
13. Karnofsky performance status < 70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Phase 1: Compare the spot to background ratio for tumor positive and tumor negative margins. | 2 years
  The main purpose is to establish the intraoperative use of cetuximab-800CW as a reliable marker for residual tumor in resection margins after surgical removal of PSCC. The objective is to establish the feasibility of cetuximab-800CW fluorescence at the dose of 75/15 mg predose/dose combination as a marker for a tumor positive resection by comparing the spot to background ratios for tumor positive and tumor negative margins. A tumor to background ratio of >2.0 is aspired.

SECONDARY OUTCOMES:
Quantification of sensitivity and positive predictive value of cetuximab-800CW in PSCC | 2 years
  To quantify sensitivity and positive predictive value of cetuximab-800CW fluorescence of PSCC ex vivo using optical molecular imaging and MDSFR/SFF versus standard immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands